CLINICAL TRIAL: NCT00364494
Title: Effect of Moderate Hemodilution During Cardiopulmonary Bypass on Postoperative Outcome Following Cardiac Surgery
Brief Title: Hemodilution and Outcome in Cardiac Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficult enrollment after the primary investigator left the centre
Sponsor: Università Vita-Salute San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DS/URC/ER/mm 556/DG
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Kidney Failure; Intraoperative Complications
Keywords: Hematocrit; Hemodilution; Blood Transfusion; Cardiopulmonary Bypass; Multiple Organ Failure; Surgery, Cardiac; Kidney Failure; Cardiac Surgical Procedures
MeSH Terms: conditions — Renal Insufficiency; Intraoperative Complications; Multiple Organ Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Different timing of red blood cells transfusion (substudy 1); Acute hemodilution versus no hemodilution (substudy 2) — Subgroup 1,with Ht<21% receive an hemotransfusion before or after CEC;subgroup 2,with Ht>25% bleed or not

SUMMARY:
An hematocrit of 21-25% is supposed to perform the best organ protection during cardiopulmonary bypass for cardiac surgery.

The investigators want to establish the best timing for a transfusion (in patients with a predicted low hematocrit during cardiopulmonary bypass) and the efficacy of preprocedural hemodilution (in patients with a predicted high hematocrit during cardiopulmonary bypass) in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiac surgery

Exclusion Criteria:

* Age < 18 years old
* Not signing written consent
* Age < 65 years old (subgroup 1)
* Emergency, aortic stenosis, main left coronary stenosis (subgroup 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
renal function

SECONDARY OUTCOMES:
other organ damage
prolonged mechanical ventilation, Intensive Care Unit (ICU) and hospital stay
sepsis
exitus

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Landoni, MD, Study Director — Università Vita-Salute San Raffaele, Milano, Italia e Istituto Scientifico San Raffaele, Milano, Italia; Giuseppe Crescenzi, MD, Principal Investigator — Università Vita-Salute San Raffaele, Milano, Italia e Istituto Scientifico San Raffaele, Milano, Italia
Locations (1):
- Università Vita-Salute San Raffaele, Milano, Italia e Istituto Scientifico San Raffaele, Milano, Italia, Milan, Italy